CLINICAL TRIAL: NCT06795152
Title: Rare Glycogen Storage Diseases Natural History Study
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00115144
Record Dates: First submitted 2025-01-22; First posted 2025-01-27 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Glycogen Storage Disease; GSD Type 0A; GSD Type 0B; GSD VII; Tarui Disease; GSD X; GSD XII; GSD XIII; GSD XV; PGBM2; PRKAG2; Danon Disease; Polyglucosan Body Myopathy Type 1; Polyglucosan Body Myopathy Type 2; RBCK1 Deficiency
Keywords: glycogen storage disease; GSD; Tarui disease; Polyglucosan Body Myopathy Type 2; PGBM2; PRKAG2; Danon disease; Polyglucosan Body Myopathy Type 1; RBCK1
MeSH Terms: conditions — Glycogen Storage Disease; Glycogen Storage Disease Type VII; Dimauro disease; Glycogen Storage Disease XII; Glycogen Storage Disease XIII; Glycogen Storage Disease Type IIb

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rare GSD (Glycogen Storage Disease): individuals with confirmed diagnosis of rare glycogen storage disease including but not limited to, GSD types 0a, 0b, VII, X, XII, XIII, XV, PRKAG2 syndrome and Danon disease
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational. Natural history study.

SUMMARY:
The purpose of this study is to collect and study key medical data about several ultra-rare GSDs (Glycogen Storage Diseases) including, but not limited to, GSD types 0a, 0b, VII, X, XII, XIII, XV, PRKAG2 syndrome and Danon disease.

DETAILED DESCRIPTION:
The immediate goal of this research is to create a natural history database to collect information from individuals who have a rare GSD. A repository of clinical, laboratory, and biochemical information on individuals with a rare GSD will allow a more definitive description of the different subtypes to be developed, which will permit development of treatment strategies in the future.

Duke will be the only site where this study takes place. However, since these are rare disorders, participants who receive care at other institutions will be included. The investigators will collect retrospective data from patient charts on diagnosed individuals, as far back as necessary to capture the clinical course of their disorder. Prospective data collected from patient charts after enrollment will be captured as well. Participant's medical records will be continually reviewed for the duration of the study.

Data will be collected from medical records and will only pertain to clinically relevant information, including, but not limited to: demographic and diagnostic information, tissue biopsy results, medical and family history, review of systems, imaging studies, results of liver, muscle, and nerve function testing, and urine and blood laboratory results.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a rare GSD, including 0a, 0b, VII, X, XII, XIII, XV, PRKAG2 syndrome or Danon disease

  * Two variants in the gene associated with the specific GSD type (for autosomal recessive diseases)
  * One variant in the gene associated with the specific GSD type (for autosomal dominant or X-linked diseases)
  * Deficient enzyme activity in liver, muscle, skin fibroblast or other tissue
  * One variant in causative gene with evidence of disease, per a clinician
  * Histology as confirmed by a clinician
* Able to provide informed consent for self (adults) or affected individual (minor or adults with a legally authorized representative)
* Able to provide consent for release of medical records
* Pregnant women with a diagnosis of a rare GSD will be included

Exclusion Criteria:

* Unable to provide informed consent for participation for one's self or by legally authorized representative/legal guardian/parent

Ages: 0 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with rare GSD, including 0a, 0b, VII, X, XII, XIII, XV, PRKAG2 syndrome and Danon disease regardless of gender or ethnicity, are eligible for enrollment
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2034-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Progression of disease confirmed by medical record review | through study completion, an average of 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Priya Kishnani, M.D., Principal Investigator — Duke
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No